CLINICAL TRIAL: NCT07039396
Title: Evaluating the Efficacy and Safety of NeoThelium FT Amnion Skin Graft in the Management of Diabetic Foot Ulcers: A Prospective Case Series
Brief Title: Prospective Case Series Evaluating the Efficacy and Safety of NeoThelium FT for Diabetic Foot Ulcers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NuScience Medical Biologics, LLC (Industry)
Collaborators: SygNola, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NeoDia
Record Dates: First submitted 2025-06-18; First posted 2025-06-26 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Diabetic Foot Ulcer
Keywords: Chronic Wounds; Cellular, Acellular, Matrix-like product (CAMP); Cellular and/or Tissue Product (CTP); Dehydrated Complete Human Placental Membrane (dCHPM)
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Intervention Model Description: NeoThelium FT in addition to Standard of Care
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NeoThelium FT + SOC (Experimental): Wound cleansing, sharps debridement, NeoThelium FT application, Dressing for moisture balance, Offloading
  Interventions: Other: NeoThelium FT (HCT/P 361)

INTERVENTIONS:
Other: NeoThelium FT (HCT/P 361) — NeoThelium FT (HCT/P 361) is a dehydrated wound covering derived from donated human placental tissue. NeoThelium FT is a dual-layer membrane with amnion and chorion combination layers.

SUMMARY:
This is a prospective case series evaluating the efficacy and safety of NeoThelium FT Amnion Skin Graft in the Mangement of Diabetic Foot Ulcers

DETAILED DESCRIPTION:
This research will take place across multiple medical centers, where both researchers and participants will know which treatment is being used (open label). Patients who agree to participate and meet the study requirements during screening will begin SOC plus NeoThelium FT weekly applications. The subject will continue follow-up per the original schedule. As this is a post-marketing study, it will gather information regarding the efficacy of treatment while also supporting insurance reimbursement decisions.

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female, 18 years of age or older
2. Subject has a medical diagnosis of Type I or Type II Diabetes Mellitus requiring oral or glycemic control and/or insulin replacement therapy with a diabetic foot ulcer
3. Subject has a diabetic foot ulcer of Wagner grade 1, 2, or 3 without infection or clinically visible exposed bone. Wagner 3 is acceptable if the diagnosis is acute osteomyelitis and the subject has successfully completed IV antibiotic treatment prior to screening.
4. Ulcer area is a minimum of 0.5 cm2 and a maximum of 25 cm2 at first treatment visit
5. Subject is able and willing to follow the protocol requirements
6. Subject had signed informed consent
7. Adequate circulation if wound is location on the lower extremity demonstrated by an ABI of >0.7 and <1.3, or TBI of >0.6 within 30 days prior to informed consent OR an arterial ultrasound noted with patent circulation and without significant stenosis 90 days prior to the first treatment visit.
8. Diabetic foot ulcer is being treated with TCC offloading therapy OR Fixed Ankle Walker if approved by Medical Monitor for 7 days prior to treatment visit 1
9. Wound free of clinical infection (no purulent discharge, cellulitis, or osteomyelitis) post-debridement.
10. Record of serum hemoglobin A1c within 90 days prior to the first treatment visit

Exclusion Criteria:

1. Subject is unable to comply with protocol treatment
2. Target ulcer is a Wagner 3 of acute osteomyelitis that has not been successfully treated with 6 weeks of IV antibiotics or is diagnosed as chronic refractory osteomyelitis.
3. Wagner 3, 4, or 5 involving tendon, bone, or joint.
4. Presence of systemic infection, sepsis, or osteomyelitis at screening.
5. Multiple DFUs on the same foot with < 2 cm separation from the target ulcer.
6. Subject has major uncontrolled medical disorders in the opinion of the investigator, such as serious cardiovascular, renal, liver, pulmonary, autoimmune, palliative care, or inherited blood disorders that may affect wound healing.
7. Subject actively being treated for malignant disease or history of malignancy or radiation therapy at the site of wound.
8. Subject has comorbid conditions that may compromise subject safety in the opinion of the investigator
9. Known contraindications or hypersensitivity to amniotic membrane products or components of NeoThelium FT.
10. Concurrent participation in alternative clinical trial that involves investigational drug or HCT/P interfering with wound treatment and/or healing.
11. Subject is pregnant or breastfeeding
12. Subject with history of immunosuppressant treatment (systemic corticosteroids >10mg daily dose), cytotoxic chemotherapy, or topical steroid application to the ulcer surface for >2 weeks duration within 30 days prior to the first treatment visit; or anticipated use of the above during the course of the study
13. Wound previously treated with CAMPs, tissue engineered, or scaffold materials within 30 days prior to enrollment
14. Index ulcer suspicious of neoplasm in the opinion of the principal investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-08-26 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Complete wound closure | 1-12 weeks
  The primary endpoint will be the percentage of target ulcers that achieve complete wound closure by manual measurement utilizing a ruler.

SECONDARY OUTCOMES:
Percentage Wound Area Change | 1-12 weeks
  The percentage change in wound area from TV-1 to TV-13 will be measured weekly using standardized method of wound area measurement and physical examination.
Follow-Up Closure | 2 weeks
  Number of wounds remaining closed during the 2-week follow-up
Time to Closure | 1-12 weeks
  Average number of grafts/weeks used to achieve wound closure
Hemoglobin A1c | 1 week
  Average Sample of HbA1c

CONTACTS AND LOCATIONS:
Overall Officials: Angelina Ferguson, DNP, Study Chair — SygNola, LLC
Locations (2):
- United States (2):
  - MedCentris of Alexandria, Alexandria, Louisiana
  - MedCentris of Leesville, Leesville, Louisiana

IPD SHARING:
Plan to Share IPD: No